CLINICAL TRIAL: NCT05653375
Title: The Effect of A Mindfulness-Based Psychoeducation Program Applied With Distance Education on the Psychological Well-Being, Emotional Intelligence and Stress Levels of Youth: A Randomized Controlled Study
Brief Title: The Effects of Mindfulness-based Psychoeducation Program on Young People
Acronym: MBPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Şenay Öztürk, Assistant Professor, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/01-11
Record Dates: First submitted 2022-12-06; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Stress; Emotional Intelligence; Nursing; Psychological Well-being; Mindfulness
Keywords: Minfulness; stress; emotional intelligence; psychological well-being; nursing
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mindfulness-based psychoeducation program (Experimental): The group in which the mindfulness-based psychoeducation program was applied.
  Interventions: Other: Mindfulness-based psychoeducation program
- control group (Active Comparator): The group in which no intervention was made and only the pre-test and post-test were applied for comparison.
  Interventions: Other: ongoing life

INTERVENTIONS:
Other: Mindfulness-based psychoeducation program — In this study, a mindfulness-based psychoeducation program was applied to the experimental group, 2 times a week for 4 weeks, with a total of 8 sessions, including methods such as meditation, body scanning, mindful eating, and breathing work. Measurement tools were applied to the experimental and control groups before and after the program.
  Arms: mindfulness-based psychoeducation program
Other: ongoing life — The control group continued with their lives without any intervention. Only pre-test and post-test were applied. While the program was applied to the experimental group, no intervention was made to the control group.
  Arms: control group

SUMMARY:
Purpose: The fact that young people starting university during the pandemic period continue this academic period with distance education increases the stress they experience. Therefore, the purpose of this study is to determine the effect of mindfulness-based psychoeducation program applied with distance education on the psychological well-being, emotional intelligence, and stress levels of youth.

Method: This study was conducted in a randomized controlled manner with a pretest-posttest control group random design model. The population of the study consisted of 120 newly enrolled students in the nursing department of a foundation university, and the sample consisted of a total of 59 students who met the inclusion criteria of the study. In the sample, while 29 students formed the intervention group, 30 students formed the control group. Mindfulness-Based Psychoeducation Program (MBPP) was applied to the intervention group twice a week for 4 weeks. Perceived Stress Scale (PSS-14), Psychological Well-Being Scale (PWB), and Revised Schutte Emotional Intelligence Scale (SEIS) were used as measurement tools. Further, t-test, Mann Whitney U analysis, and Wilcoxon signed-row test were used in the analysis of the data.

DETAILED DESCRIPTION:
Population-Sample: The population of this study consisted of 1st grade students registered at Maltepe University School of Nursing in the 2020-2021 academic year. 64 students who met the criteria for participating in the study (over 18 years of age, without a psychiatric diagnosis, who did not practice mindfulness before, who did not meditate, whose mother tongue was Turkish, who scored above the cut-off point (25˂) in the perceived stress scale) and declared their willingness to be a voluntary participant formed the sample. G*Power 3.1.9.2 program was used to estimate the number of samples (Faul, Erdfelder, Lang et al. (2007). In order to calculate the effect size in power analysis, the relevant literature was examined and the study by Yılmaz (2021) was taken as a basis. The effect size value (Cohen's d) calculated with the emotional intelligence score averages and standard deviations (intervention group= 92.73 ± 13.01; control group = 81.80 ± 8.95) of the intervention and control groups presented in Yılmaz's (2021) study was calculated as .98. In this study, it was determined that, for the one-tailed hypothesis, the minimum number of samples to be included in the study with an effect size of .98, a margin of error of 0.05, and a power of 0.95 should be 48 people in total, 24 for each group (intervention group = 24; control group = 24). Participants were numbered from 1 to 64, and 32 intervention and 32 control groups were created from the www.random.org site, taking into account the possibility of data loss. During the application process, 2 people from the intervention group did not want to continue after the first session, 1 person had long-term internet connection problems, and 2 people from the control group did not fill out the second measurement forms (drop out). The study was completed as 29 intervention and 30 control groups.

Data collection and program application:

Before starting the research, the ethics committee decision dated 08/01/2021 and numbered 2021/01-11 was taken from X Ethics Committee. Data were collected online via google forms. On the first day of the application, other scales except the Perceived Stress Scale were applied simultaneously to the intervention and control groups. The intervention group was given a program for 4 weeks, with 2 sessions per week and each session 90 minutes. At the end of the program, data collection tools were applied to both groups simultaneously again. During this period, no application was made to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Without a psychiatric diagnosis,
* Have not done awareness practices before,
* Not meditating,
* Not a foreign national,
* Those who score moderately and above on the Perceived Stress Scale
* Those who volunteered to participate in the study

Exclusion Criteria:

* Those who scored less than 25 on the perceived stress scale.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change of psychological well-being after 4 weeks. | baseline and 4 weeks.
  Psychological Well-Being Scale: The items of the Psychological Well-Being Scale are answered between 1 and 7, as strongly disagree (1) to strongly agree (7). Scores range from 8 to 56. A high score indicates that the person has many psychological resources and strengths.
Change of emotional intelligence level after 4 weeks. | baseline and 4 weeks.
  Revised Schutte Emotional Intelligence Scale: The scale, which was studied using the total score, has three sub-dimensions and consists of 41 items. It is a Likert-type scale with items scored between 1 and 5 (1: Never, 5: Always). If the total score of the scale is high, it means that the level of emotional intelligence is also high.
Change of perceived stress level after 4 weeks. | baseline and 4 weeks.
  Perceived Stress Scale: Consisting of 14 items in total, PSS-14 is designed to measure how stressful situations in a person's life are perceived. The scores of the PSS-14 vary between 0 and 56, and the high score indicates a high perception of stress (cut-off point > 25).

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozturk S. The effect of a distance-delivered mindfulness-based psychoeducation program on the psychological well-being, emotional intelligence and stress levels of nursing students in Turkey: a randomized controlled study. Health Educ Res. 2023 Dec 11;38(6):575-586. doi: 10.1093/her/cyad040. PMID 37885327